CLINICAL TRIAL: NCT05676788
Title: Hyperspectral Imaging for Intersegmental Plane Identification During Sublobar Pulmonary Resections in Lung Cancer Patients
Brief Title: HSI for Intersegmental Plane Identification During Sublobar Pulmonary Resections
Acronym: HYPER-Seg
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: LungenClinic Grosshansdorf (Other)
Collaborators: Institute of Medical Technology and Intelligent Systems, Hamburg University of Technology, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSI_01
Record Dates: First submitted 2022-11-26; First posted 2023-01-09 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Lung Neoplasm; Pulmonary Metastasis
Keywords: Hyperspectral Imaging; Lung cancer; Segmentectomy; Indocyanine green; Intersegmental plane; Machine learning strategies
MeSH Terms: conditions — Lung Neoplasms | interventions — Hyperspectral Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intersegmental plane identification by HSI and ICG (Experimental): Hyperspectral Imaging Intersegmental plane identification:
  Defined as distance between intersegmental plane identification with Hyperspectral Imaging compared to near-infrared indocyanine green fluorescence.
  Interventions: Device: Hyperspectral Imaging

INTERVENTIONS:
Device: Hyperspectral Imaging — Identification of the intersegmental plane

SUMMARY:
The purpose of this study is the identification of the intersegmental plane and navigation during sublobar pulmonary resections in lung cancer using Hyperspectral Imaging, the comparison with ICG fluorescence intersegmental plane identification, and the establishment of automatic intersegmental plane navigation using machine learning strategies for intraoperative navigation.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer-related death worldwide. Due to the generalization of screening strategies, especially for risk populations, an increasing number of lung cancer cases are detected in an early stage. In this regard, lung cancer is also increasingly diagnosed in patients with impaired pulmonary function. For preserving lung function and reducing complication incidence, pulmonary segmentectomies are currently evaluated in this cohort. Thus, the latest version of the German guideline for the prevention, diagnosis, treatment and follow-up of lung cancer recommends segmentectomy for patients with impaired pulmonary function in tumor stage I/II. However, the identification of the intersegmental plane - the key step of segmentectomy - remains challenging. Inaccurate recognition of the intersegmental plane may lead to dysfunction of the remaining lung tissue, mismatching of ventilation or blood flow, or long-term air leakage after surgery, which even requires unplanned secondary surgery. Indocyanine green (ICG) is one the latest evaluated identification methods and is considered as gold standard. Hyperspectral Imaging (HSI) - a newly established intraoperative imaging technique - enables a non-invasive evaluation of tissue perfusion and the discrimination of pulmonary tissue with different tissue perfusion during segmentectomies.

The purpose of this prospective, single-center, non-inferiority IDEAL Stage 2b study is the identification of the intersegmental plane and navigation during sublobar pulmonary resections in lung cancer using Hyperspectral Imaging, the comparison with ICG fluorescence intersegmental plane identification, and the establishment of automatic intersegmental plane navigation using machine learning strategies for intraoperative navigation.

To address this, the intersegmental plane will be detected by both HSI and ICG-fluorescence during pulmonary segmentectomies and the correspondence of the two identification methods will be compared with one another. Using machine learning strategies, the detection of perfused and non-perfused pulmonary tissue and intersegmental plane will be analyzed. Finally, the investigators will study motion tracking for the improvement of future HSI illustrations during surgery.

The hypothesis of this study is that HSI could improve the intraoperative navigation during pulmonary segmentectomies providing as reliable intersegmental plane identification as the gold standard of indocyanine green fluorescence. In this case, an intravenous application of fluorescent dye would not be required anymore for the intersegmental plane identification.

In the case of complex segment resection, a large amount or repeated use of ICG is necessary due to its short pulmonary circulation time. Multiple use of ICG may result in ICG entering the target lung tissue through the bronchial circulation and increases the risk of adverse drug reactions of ICG. In contrast, the advantages of HSI would be a faster and repetitive measurement during surgery. There will be a potential for reducing the total measurement time during intersegmental plane dissection (10 seconds vs. 3 minutes / measurement) and consequently patient's burden. In this context, several studies of HSI-based perfusion measurement during esophageal or colorectal surgery showed already an improved patients' outcome. Furthermore, HSI can be used for surgery on patients with hyperthyroidism or impaired renal or hepatic function.

In order to support this hypothesis, a prospective non-inferiority trial design will be used in this study. To ensure the quality of data acquisition and reporting, the study will be conducted in accordance with the IDEAL reporting guidelines. During pulmonary segmentectomies, the intersegmental plane will be identified by both HSI and ICG fluorescence. The determined HSI intersegmental margin will be benchmarked against the ground truth ICG fluorescence and the feasibility and reproducibility of HSI and ICG mapping will be studied.

Machine learning methods have greatly improved the interpretation of subtle patterns in medical image data. Convolutional neural networks (CNNs) can be considered state-of-the-art for classification and segmentation of medical images. The investigators will extend CNN-based methods for HSI classification and particularly study patch-based differentiation between perfused and non-perfused tissue using ICG and HSI data acquired at the same position. A further challenge is the relatively slow acquisition of HSI (10 seconds/measurement), which makes it prone to motion artifacts, e.g., due to pulsatile motion. To address this, the investigators will study motion tracking, which is also relevant for the future illustration of the segment boundary during surgery.

Machine learning approaches and particularly CNNs allow to directly optimize classifiers based on actual clinical data and the spectral dimension can be handled in a straightforward fashion. Moreover, as a versatile method for image processing, CNNs can also be used for localization and motion compensation during intraoperative imaging, e.g., they can be trained to detect image features and their motion in red/green/blue image streams. This is interesting for the proposed HSI data acquisition, which is based on a sequence of measurements which are sensitive to tissue motion.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed lung cancer stage I/II or malignancy suspicious nodules
2. Segmentectomy is oncologically indicated or impaired pulmonary and/or cardiac function prevent anatomical resection
3. Male or female patients aged ≥ 18 years without upper age limit
4. Serum creatinine ≤ 1.5 x upper limit of normal or creatinine clearance (CrCl ≥ 50 mL/min, Cockcroft-Gault formula)
5. Total bilirubin ≤ 1.5 x upper limit of normal (except patients with Gilbert Syndrome (Morbus Meulengracht) in whom total bilirubin < 3.0 mg/dL is allowed)
6. Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase)/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase) ≤ 2.5 x upper limit of normal
7. Full legal capacity
8. Written informed consent obtained according to international guidelines and local laws
9. Ability to understand the nature of the trial and the trial related procedures and to comply with them

Exclusion Criteria:

1. Requirement of a lobectomy or pneumonectomy to achieve complete resection
2. Allergy to indocyanine green or iodine
3. Hyperthyroidism
4. Current or planned pregnancy, nursing period (if defined as requirement of clinical routine treatment)
5. Medical condition which poses a high risk to undergo surgery as defined by the investigator
6. Covid19 / SARS-CoV2-infection at time of screening
7. Participation in any other interventional clinical trial within the last 30 days before the start of this trial
8. Simultaneous participation in other interventional trials which could interfere with this trial; simultaneous participation in registry and diagnostic trials is allowed
9. Known or persistent abuse of medication, drugs or alcohol
10. Person who is in a relationship of dependence/employment with the coordinating investigator or the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Intersegmental Plane identification | directly before pulmonary intersegmental plane dissection
  Distance between intersegmental plane identification with Hyperspectral Imaging compared to near-infrared indocyanine green fluorescence

SECONDARY OUTCOMES:
Tumor distance [mm] | immediately after surgery
  Shortest distance between tumor and HSI and ICG-fluorescence predicted intersegmental plane
7-item binary rating scale for feasibilty of HSI measurement | immediately after surgery
  Evaluation of feasibility of HSI and ICG-fluorescence intersegmental plane identification using a 7-item binary rating scale

OTHER OUTCOMES:
Machine Learning | one week after surgery
  Intersegmental plane identification with machine learning strategies. To predicted intersegmental plane by the machine learning algorithm developed in this project. The machine learning algorithm is trained on thoracoscopic HSI image and specimen data to predict if the intersegmental plane is displayed correctly during surgery.
Safety of HSI | at 10 days and 6 weeks after surgery
  Safety will be evaluated by measuring the rates of adverse reactions to HSI and ICG dye, intraoperative complications, and perioperative complications using the Ottawa Thoracic Morbidity and Mortality Classification

CONTACTS AND LOCATIONS:
Locations (1):
- LungenClinic Großhansdorf, Großhansdorf, Germany